CLINICAL TRIAL: NCT02978391
Title: A Prospective, Multicenter, Single-blind, Controlled Clinical Trial to Confirm the Efficacy and Safety of 'UI-EWD', a Wound Dressing Used for Wound Protection and Hemostasis After Ulcer Bleeding Due to Peptic Ulcer, EMR and ESD
Brief Title: UI-EWD for Endoscopic Hemostasis of Bleeding Peptic Ulcers and Bleeding After EMR/ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEXTBIO-631-EWD3
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2017-09

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- UI-EWD Hemostatic system (Experimental): Patients with upper gastrointestinal bleeding treated with UI-EWD
  Interventions: Device: UI-EWD Hemostatic system
- epinephrine (Active Comparator): Patients with upper gastrointestinal bleeding treated with submucosal epinephrine injection
  Interventions: Drug: epinephrine endoscopic injection (conventional therapy)

INTERVENTIONS:
Device: UI-EWD Hemostatic system — Adhesive endoscopic hemostats, powder type
  Arms: UI-EWD Hemostatic system
Drug: epinephrine endoscopic injection (conventional therapy) — endoscopic submucosal injection of epinephrine (1: 10,000)
  Arms: epinephrine

SUMMARY:
UI-EWD (NextBiomedical Co, Incheon, South Korea), a new hemostatic powder for endoscopic treatment of high-risk bleeding peptic ulcers and bleeding after ESD/EMR.

DETAILED DESCRIPTION:
UI-EWD (Endoscopic Wound Dressing) is adhesive absorbable powder as a new hemostasis material, the therapeutic effect and safety in endoscopic application will be verified. This study has been designed to observe comparing UI-EWD versus the submucosal epinephrine injection for endoscopic hemostasis of bleeding peptic ulcers and bleeding after EMR/ESD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bleeding peptic ulcer and active bleeding after ESD/EMR

Exclusion Criteria:

* Coagulation disorder (PLT < 50*10^9/L, INR > 2)
* Connot stop taking the antiplatelet drug, NSAID, Anticoagulant drug, and Aspirin during endoscopic treatment and after 72h endoscopy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Recurrent bleeding rate | 3 days
  Rebleeding rate up to 3 days was obtained by clinical manifestations such as melana; decreased hemoglobin > 2g/dL; hemodynamic instability or active bleeding from mucosal defect under endoscope.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Woon Shin, Principal Investigator — Inha University Hospital
Locations (2):
- South Korea (2):
  - Soonchunhyang University College of Medicine, Bucheon-si
  - Inha University Hospital, Incheon